CLINICAL TRIAL: NCT04289467
Title: A Phase II Study of Fenfluramine for Treatment of Refractory Infantile Spasms
Brief Title: Treatment of Refractory Infantile Spasms With Fenfluramine
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Orange County (Other)
Responsible Party: Principal Investigator, Daniel Shrey, Associate Professor, Children's Hospital of Orange County
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZX008-IS
Record Dates: First submitted 2020-02-21; First posted 2020-02-28 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Infantile Spasm
MeSH Terms: conditions — Spasms, Infantile | interventions — Fenfluramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fenfluramine treatment (Experimental): Open label treatment with fenfluramine. Dosage will be titrated to 0.8 mg/kg/day, for an initial duration of 21 days. Patients with favorable response will have an option to continue treatment for up to 6 months.
  Interventions: Drug: Fenfluramine

INTERVENTIONS:
Drug: Fenfluramine — Open-label
  Other Names: Fenfluramine Hydrochloride

SUMMARY:
This is a phase II clinical trial in which children with refractory infantile spasms (also called epileptic spasms or West syndrome) will be treated with fenfluramine, to evaluate efficacy, safety, and tolerability. Patients with infantile spasms that have not responded to treatment with vigabatrin and ACTH we will be invited to participate. Study participants will undergo baseline video-EEG, receive treatment with fenfluramine for 21 days, and then undergo repeat video-EEG to determine effectiveness. Patients with favorable response will have the opportunity to continue treatment for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 12 to 36 months, inclusive
* Clinical diagnosis of infantile spasms
* Continued epileptic spasms despite adequate treatment with ACTH and vigabatrin.

Exclusion Criteria:

* Significant preexisting cardiovascular disease
* Exposure to any cannabinoid product within 14 days of screening
* Initiation or dose-titration of any second-line treatment for infantile spasms in the 14 days prior to screening.
* Implantation of a vagal nerve simulator within 14 days of screening
* Initiation and maintenance of the ketogenic diet within 3 months of screening

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Electroclinical response (Efficacy) | 12 months
  Number of participants with resolution of epileptic spasms and hypsarrhythmia (if present at baseline) after 21 days of treatment, as determined by overnight video-electroencephalography (EEG) evaluation and caregiver seizure diary.

SECONDARY OUTCOMES:
Computational electroencephalography response (Efficacy) | 12 months
  Median and range of response quantified using the probability-weighted response index (PWRI), a novel computational electroencephalography measure of hypsarrhythmia burden.
Incidence of treatment emergent adverse events (Safety and tolerability) | 12 months
  Detailed accounting of all treatment-emergent adverse events, including number of participants with clinically-significant valvulopathy and/or pulmonary hypertension, as determined by echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Shrey, MD, Principal Investigator — Children's Hospital of Orange County
Locations (2):
- United States (2):
  - UCLA Health, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California

IPD SHARING:
Plan to Share IPD: No